CLINICAL TRIAL: NCT05509010
Title: AI Driven National Platform for CT cOronary Angiography for clinicaL and industriaL applicatiOns Registry (APOLLO)
Brief Title: AI Driven National Platform for CT cOronary Angiography for clinicaL and industriaL applicatiOns Registry
Acronym: APOLLO
Status: Recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Other Study IDs: APOLLO
Record Dates: First submitted 2022-04-19; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: CAD; Coronary Artery Disease; Coronary Stenosis; Plaques; Epicardial
Keywords: CTCA; CT Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Plaque, Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: 4000 patients who were clinically evaluated by CTCA from 1 Jan 2007 to 31 Oct 2017.
  Interventions: Procedure: CTCA
- Prospective: 4000 patients who are clinically evaluated by CTCA.
  Interventions: Procedure: CTCA

INTERVENTIONS:
Procedure: CTCA — CTCA is performed as part of routine care procedure.

SUMMARY:
The overall aim is to build an AI driven national Platform for CT cOronary angiography for clinicaL and industriaL applicatiOns (APOLLO) for automated anonymization, reporting, Agatston scoring and plaque quantification in CAD. It is a "one-stop" platform spanning diagnosis to clinical management and prognosis, and aid in predicting pharmacotherapy response.

DETAILED DESCRIPTION:
Coronary artery disease (CAD), a blockage of the blood vessels, affects 6% of the general population and up to 20% of those over 65 years of age. CAD is a leading cause of cardiac mortality in Singapore and worldwide, with 19% of deaths in Singapore due to CAD (MOH website).

Numbers of CAD cases are increasing due to ageing and the higher prevalence of contributary diseases such as diabetes. Computed Tomography Coronary Angiography (CTCA) is the first-line investigation for CAD as indicated by the National Institute for Clinical Excellence (NICE) guidelines. Recent Prospective Multicenter Imaging Study for Evaluation of Chest Pain (PROMISE) and Scottish Computed Tomography of the Heart (SCOT-HEART) trials support CTCA as the dominant means for evaluating coronary anatomy and physiology as it increases diagnostic certainty, improves efficiency of triage to invasive catheterization and reduces radiation exposure when compared to functional stress testing.

Currently, CAD report generation requires 3-6 hours of a CT specialist's time to annotate scans, with inter-observer variability of 20%. In addition, there is no effective singular toolkit to analyse Agatston scores (a measure of calcified CAD), severity of stenosis, and plaque characterisation.

These problems have severely constrained the effectiveness of CTCA as a diagnostic and research tool. The investigators plan to build upon Singapore's competitive advantages in artificial intelligence (AI) to provide a solution to these gaps.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years old
2. Signed informed consent
3. Clinically indicated for evaluation by CTCA

Exclusion Criteria:

1. Individuals unable to provide informed consent
2. Known complex congenital heart disease
3. Planned invasive angiography for reasons other than CAD
4. Non-cardiac illness with life expectancy < 2 years
5. Pregnancy
6. Concomitant participation in another clinical trial in which subject is subject to investigational drug or device
7. Cardiac event and/or coronary revascularization (percutaneous coronary intervention (PCI) and/or coronary artery bypass grafting (CABG) and/or valvular repair/replacement prior to CTCA
8. Glomerular Filtration Rate ≤ 30mL/min
9. Known allergy to iodinated contrast agent
10. Contraindications to beta blockers or nitroglycerin or adenosine

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are clinically evaluated by CTCA
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
AI precision toolkits: AI stenosis reporting | baseline
  Stenosis reporting: Severity of stenosis and accurate anatomical localization of stenosis.
  The significance of a stenosis is determined by visual estimation of the maximal grade of luminal narrowing caused by the plaque. As recommended in SCCT guideline (Leipsic et al., 2014) , coronary stenosis can be graded as minimal, mild, moderate, severe and total occluded separately. Following the guideline, a stenosis will be classified as obstructive and non-obstructive. The location of the stenosis uses the SCCT model (Leipsic et al., 2014)
AI precision toolkits: Agatston scoring | baseline
  Agatston scoring: Agatston scoring of calcified plaque. As recommended in SCCT clinical practical guidelines (Leipsic et al., 2014), Agatston scoring programs generally identify pixels that exceed 130 HU as a level corresponding to calcium on a non-contrast study (Agatston et al., 1990) . The reader needs to identify each lesion discrete calcific focus) in each vessel distribution. The summed score for each vessel is generated by the scoring program based on an area-density (Agatston score) (Agatston et al., 1990) measurement of each calcified focus. The total coronary Agatston score is the sum of all calcified lesions in all coronary beds.
AI precision toolkits: Plaque | baseline
  Plaque analysis: Plaque volume, burden, type and anatomical locations. Coronary segmentation and plaque analysis is performed for segments with diameter ≥1.5 mm. Location of plaque uses the SCCT model (Leipsic et al., 2014). For each plaque, the reader marks its start-and end-points, quantifies plaque area,volume and plaque burden, and specifies its type (non-calcified, calcified, or mixed) (Achenbach et al., 2004) . Additionally, non-calcified plaque can be further divided into low attenuation plaque (LAP). A HU <30 will signify LAP and >30 will signify non-LAP.
AI precision toolkits: EAT analysis | baseline
  EAT analysis: Total volume and anatomical locations. EAT and pericardial adipose tissue (PAT) are metabolically active fat surrounding the coronary artery and the heart, being associated with increased risk of cardiovascular disease (Villasante et al, 2019) . EAT can be quantified on non-contrast CT scans. The annotations on the CT scans are obtained by manually drawing the pericardium first to define the region. EAT is identiﬁed using the adipose tissue attenuation references between -190 and -30 HU (Oikonomou et al., 2018) . Due to the CT scan noise and changing of attenuation, the HU value of fat can vary, so the final EAT region is verified by an experienced radiologist or cardiologist.

SECONDARY OUTCOMES:
AI outcome analysis | one to five years from baseline
  1. Mortality (All-cause and/or cardiovascular)
AI outcome analysis | one to five years from baseline
  Major-adverse cardiovascular events (myocardial infarction, stroke, heart failure, revascularisation, arrhythmias, etc)
AI outcome analysis | one to five years from baseline
  Re-hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Liang Zhong, Principal Investigator — National Heart Centre Singapore
Locations (3):
- Singapore (3):
  - National Heart Centre Singapore, Singapore
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leng S, Cheng N, Tan E, Baskaran L, Teo L, Yew MS, Ngiam KY, Huang W, Chai P, Ong CC, Sia CH, Singh M, Loong YT, Raffiee NAS, Wang X, Allen J, Tan SY, Chan M, Lee HK, Zhong L. Deep learning-based quantification of epicardial adipose tissue volume from non-contrast computed tomography images: a multi-centre study. Eur Heart J Digit Health. 2025 Oct 13;6(6):1223-1233. doi: 10.1093/ehjdh/ztaf116. eCollection 2025 Nov. PMID 41267847
- [Derived] Baskaran L, Leng S, Dutta U, Teo L, Yew MS, Sia CH, Chew NW, Huang W, Lee HK, Vaughan R, Ngiam KY, Lu Z, Wang X, Tan EWP, Cheng NZY, Tan SY, Chan MY, Zhong L; APOLLO investigators. Cohort profile: AI-driven national Platform for CCTA for clinicaL and industriaL applicatiOns (APOLLO). BMJ Open. 2024 Dec 2;14(12):e089047. doi: 10.1136/bmjopen-2024-089047. PMID 39622571
- [Derived] Wang X, Leng S, Lu Z, Huang S, Lee BH, Baskaran L, Yew MS, Teo L, Chan MY, Ngiam KY, Lee HK, Zhong L, Huang W. Context-aware deep network for coronary artery stenosis classification in coronary CT angiography. Annu Int Conf IEEE Eng Med Biol Soc. 2023 Jul;2023:1-4. doi: 10.1109/EMBC40787.2023.10340650. PMID 38083399